CLINICAL TRIAL: NCT03202095
Title: Creatine for Treatment of Depression Associated With Type 2 Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No referral from diabetes clinic.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Perry Renshaw, MD, PhD, MBA, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00101803
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Type 2 Diabetes; Creatine; Diabetes
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Treatment with Creatine (Experimental): 5 grams daily of oral creatine monohydrate powde
  Interventions: Drug: Creatine Monohydrate

INTERVENTIONS:
Drug: Creatine Monohydrate — 5 grams daily of oral creatine monohydrate powder.

SUMMARY:
The investigators hypothesize that the administration of a widely available, naturally occurring dietary supplement, creatine monohydrate, will reduce the severity of depression in individuals with type 2 diabetes. The purpose of this study is to determine whether 12 weeks of creatine supplementation is an effective treatment for depression in individuals with type 2 diabetes.

DETAILED DESCRIPTION:
Depression is a debilitating illness associated with diminished quality of life and significant personal and societal costs. Depression is twice as common in those with type 2 diabetes compared to the general population. Antidepressants are commonly prescribed as treatment for depression; however, they may not be the optimal treatment for people with type 2 diabetes. Creatine has been shown to decrease symptoms of depression in many types of individuals when used over the course of 8 weeks or more. The purpose of this study is to investigate whether creatine can decrease symptoms of depression in individuals with type 2 diabetes when taken daily for 12 weeks. This study also investigates how creatine impacts brain chemistry as creatine decreases depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Major Depressive Disorder identified by the SCID-5-RV
* Current HAM-D score of > 16
* Current type 2 diabetes (as confirmed by clinical history and baseline glycosylated hemoglobin percentage (HgA1c) > 6.5.
* Diabetes type II present for at least one year

Exclusion Criteria:

* Diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder, identified by the SCID-5-RV
* History of or current diagnosis of acute kidney injury (AKI), chronic kidney disease (CKD) or end-stage renal disease (ESRD)
* Electrolyte disturbance (hypokalemia, hyperkalemia, hyponatremia, or hypernatremia) on screening basic metabolic panel
* History of cardiac disease or QTc >500ms on screening EKG
* History of diabetic ketoacidosis or hyperosmolar hyperglycemic state
* History of seizure disorder
* Current serious suicide risk identified by the Columbia Severity Suicide Rating Scale
* Positive pregnancy test
* Breastfeeding
* Contraindication to an MRI scan
* Current incarceration

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Depression Rating Scale | 12 weeks
  The purpose of this study is to determine whether 12 weeks of dietary creatine augmentation with oral 5 g creatine daily reduces hypoxia-related depressive symptoms measured by the 17-item Hamilton Depression Rating Scale (HAM-D) in women with SSRI or SNRI resistant depression.

CONTACTS AND LOCATIONS:
Overall Officials: Perry F Renshaw, MD, PhD, MBA, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No